CLINICAL TRIAL: NCT02571309
Title: Asthmatuner a Self-management App for Asthma
Brief Title: Asthmatuner a Self-management App for Asthma: A Randomized Controlled Multicentre Trial
Acronym: Asthmatuner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Björn Nordlund, PhD RN, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Medituner-001
Record Dates: First submitted 2015-09-20; First posted 2015-10-08 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Asthma
Keywords: Self-management; Asthma; Patient education; Health literacy; Health-related quality of life; Asthma control; Adherence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smartphone app - Asthmatuner (Other): The app Asthmatuner contains four different modes;
  1. Lung function testing with Bluetooth connection of external spirometry
  2. Symptom evaluation
  3. Actual treatment plan, based om lung function and symptoms
  4. Trend views of lung function, symptoms and asthma control
  Interventions: Device: Asthmatuner
- Conventional (Other): Conventional treatment and Asthmatuner will be stratified and harmonized into categories of asthma management and current state-of-art at each health care centre. Each group harmonized group will include 43 subjects.
  Interventions: Device: Asthmatuner

INTERVENTIONS:
Device: Asthmatuner — Asthmatuner is an app for self-management of asthma.

SUMMARY:
Primary aim: Evaluating the effect of Asthmatuner on patients´ self-reported asthma control test (ACT/C-ACT)compared with conventional asthma management.

Secondary aim: Evaluating patients´ health-related quality of life (HR-QoL) medical adherence by using Asthmatuner compared with conventional management.

Total sample size: Stratified study population consisting of 43 females and males with diagnosed asthma at the age of at least 6 years pediatric specialist care and 43 females/males in primary care.

Study design: This is a multi-centre, blinded, randomized controlled, cross-over trial over to at least 16 weeks.

Subjects: Two stratified groups of participants with uncontrolled asthma will be recruited; (1) children and adolescents from Astrid Lindgren's Children's Hospital, Karolinska University Hospital, and (2) adolescents and adults from the primary health care sector in Stockholm, Sweden. The asthma control test (ACT/C-ACT) will be applied for evaluation of asthma control, a score less than 20 will be required for inclusion.

Intervention: Asthmatuner is an app supporting self-management evaluating symptoms and lung function with external spirometry. The app gathers the information to define patients´ asthma control. Subsequently, Asthmatuner provides the patient with a treatment recommendation based on the individual treatment plan.

Procedures: Participants are randomized (1:1) into the one of two-arms of asthma self-management with Asthmatuner - conventional or conventional - Asthmatuner. Questionnaires will collect information about asthma control, HR-QoL, Medicine adherence report scale (MARS) and history of medical health concerning health care utilization and personal costs and income.

Analysis: The study hypothesis will be tested by examining difference in patients´ change in asthma control (ACT/C-ACT) and HR-QoL (PAQLQ/Mini-AQLQ). Results will be summarized at each management period as mean scores and analysed by paired t-tests.

DETAILED DESCRIPTION:
2. Background Clinical gaps hamper proper asthma management, and leads to delayed or undiagnosed disease, poor adherence to treatment, inadequate self-care abilities, inadequate understanding of disease severity, poor patient education, inadequate measurement of lung function, and inconsistent evaluation of symptoms. To improve the patient's ability to self-manage and to overcome clinical gaps, evidence emphasizes clinics to offer comprehensive patient education. The national Finish asthma programme (1994-2004) focused on applying effective strategies of asthma management, as a result, patient's self-management was improved, and cost-effective through limited demands on the health-care and social security system.

Novel applications embodied in smartphones are straightforward alternative to facilitate health care and support patients with hands-on guidance for self-management of asthma. Asthmatuner is a smartphone app that enables evaluation of lung function and symptoms. The app provides patients with a daily treatment plan adjusted for symptoms and lung function. Additionally, information is accessible and can be assessed by health care providers through a back-end system. Future versions of Asthmatuner will be enabled through patient's own medical record. Self-management apps with hands-on guidance for self-management of asthma present a promising future for closing clinical gaps, but the overall benefits of using the service in the treatment of asthma need comprehensive evaluation that answers scientific questions and end-user opinions.

3. Aims The primary aim is to evaluate Asthmatuner and the clinical effect on patients´ self-reported asthma control test (scores of ACT/C-ACT).

The secondary aim is to evaluate the effect on patients´ and HR-QoL and medical adherence.

Primary outcomes The primary outcome will be scores of ACT/C-ACT and Paediatric asthma quality of life questionnaire (PAQLQ) or Mini-Asthma Quality of Life Questionnaire (Mini-AQLQ).

Secondary outcomes The secondary outcomes are scores of Medicine adherence report scale (MARS) and costs of prescribed dose and type of control medication and total amount of direct and indirect costs for patient/caregiver.

4. Material and methods Study design: Multicenter randomized controlled physician blinded crossover trial, where study participants were randomized to start with AsthmaTuner or conventional treatment, and a washout period between treatments, Figure 1. Primary outcome of asthma control test (ACT) or Childhood Asthma Control Test (C-ACT) were measured two times in each treatment period, at baseline and at follow-up visit, equal or more than 8 weeks after treatment started. The participating centers were recommended to comply with Swedish national treatment and management of asthma, which closely resemble with Global Initiative for Asthma (GINA). A study nurse at each site performed the randomization by open a sealed envelope indicating the start of either AsthmaTuner or conventional treatment. The physician was blinded for the order of given treatments when one paper personalized treatment plan and one individual treatment plan for AsthmaTuner were arranged to each patient according to levels of controlled, partly controlled and uncontrolled asthma. The regional board of Ethical Committee in Stockholm (number: 2015/1527-31/1 and 2016/1546-32) and Swedish Medical Products Agency (number 5.1-2016-19829) both approved the study. The study was registered at ClinicalTrial.gov

Intervention: Asthmatuner is a CE-marked cloud-based system with healthcare interface and a downloaded patient app (Android or iOS). The intended use of Asthmatuner is to automate and facilitate self-management of asthma, by letting patient register symptoms and to measure forced expiratory volume in one second (FEV1) with a Bluetooth spirometer (MIR, SmartOne). The patient receives an immediate feedback on asthma control and treatment recommendation with an image of the correct inhaler to use and the dose. Asthma control is defined based on to GINA and a summary of lung function; liter to percentage of personalized best FEV1 using cutoff equal or less than 80%, and asthma symptoms last week in terms of; need for recue medication more than twice, daytime symptoms, nocturnal symptoms/awakenings and limitation of activities. Furthermore, Asthmatuner offers patient and asthma care provider a longitudinal data view of prescribed treatments, lung function and experienced symptoms.

Study subjects, children from 6 years and adults, with doctor's diagnosis of asthma and ACT or C-ACT score below 20 points, were included in the region of Stockholm, Sweden. The study was conducted in the primary health care sector and in asthma clinics specialised for children and adolescents in Stockholm. Patients were included at Liljeholmen Health Care Centre, Sophiahemmet Health Care Centre, and Astrid Lindgren Children's Hospital (Lung- and Allergy Department in Solna and Children and Adolescents Health Care Department in Huddinge) during the years of 2016-2018. Exclusion criteria were other ongoing comorbidity impairing the asthma control, participation in other drug trial, and a patient or all caregiver(s) (in case the patient is a child) incapable to read Swedish.

Data collection

Questionnaires:

* A health questionnaire completed at the first visit will provide information regarding asthma medical history, health utilization, annual income and employment status.
* ACT will be used to assess asthma control in patients 12 years or older, and C-ACT in children of age 6 to 11 years. A mean score equal or below 19 indicates uncontrolled asthma. Scores above 19 defines asthma to be controlled in both tests.
* HR-QoL will be applied in patients from 6 to 11 years of age using the validated Swedish translated Paediatric Asthma Quality of Life Questionnaire (PAQLQ), and the mini Asthma Quality of Life Questionnaire (mini-AQLQ) in patients from 12 years of age.
* Self-reported medication adherence will be measured with five-item MARS, developed to assess adherence with asthma medication. The MARS comprises statements about medication use behaviors. The patient is asked to answer each behavior with a score between 1-5 based on of following alternatives; "always", "often", "sometimes", "rarely" or "never". A mean MARS score will then be calculated, and a score of 4.5 or greater indicates good adherence.
* Time consume, utility and satisfaction using Asthmatuner will be asked patient/caregiver, nurses and physicians in relation to applied management.

Power analysis The power analysis is based on our previous analysis of ACT/C-ACT and HR-QoL scores in schoolchildren with uncontrolled severe asthma [21]. The scores for severe uncontrolled asthma were on average for ACT 17 (SD 3.3) and for PAQLQ 5.4 (SD 0.77). Thus, an estimated improvement of ACT from 17 to 19 (two points) or PAQLQ from 5.4 to 5.9 (0.5 points) requires 38-43 patients in each group (Asthmatuner vs. conventional management) to attain an 80 % power at 5% significance level.

Visit 1: Eligibility of participants will be checked. The patient will be given information about the study procedures and must sign the informed consent form. At the visit the following procedures will be conducted and documented:

* Demographic data
* Body height and weight
* Medical history about allergy and asthma will be obtained with health questionnaire
* Asthma control will be assessed with ACT or C-ACT
* HR-QoL; Mini-AQLQ or PAQLQ
* MARS questionnaire
* Lung function, dynamic spirometry including forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC, forced expiratory flow after 50% of vital capacity (FEF50)
* Randomization to; Asthmatuner - conventional self-management or conventional - Asthmatuner
* Prescribe and apply treatment plan (Asthmatuner or Conventional)
* Control of inhalation technique

At visit 2, the following procedures will be conducted and documented:

* ACT/C-ACT
* HR-QoL; Mini-AQLQ/PAQLQ
* MARS
* Lung function, dynamic spirometry (FVC, FEV1, FEV1/FVC and FEF50)
* Revise treatment plan if necessary (Asthmatuner or Conventional)
* Revision of adverse events.

At visit 3, the following procedures will be conducted and documented:

* ACT/C-ACT
* HR-QoL; Mini-AQLQ/PAQLQ
* MARS
* Lung function, dynamic spirometry (FVC, FEV1, FEV1/FVC and FEF50)
* Prescribe and apply treatment plan (Asthmatuner or Conventional)
* Control of inhalation technique
* Revision of adverse events.

At visit 4, the following procedures will be conducted and documented:

* ACT/C-ACT
* HR-QoL; Mini-AQLQ or PAQLQ
* MARS
* Lung function, dynamic spirometry including forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC, forced expiratory flow after 50% of vital capacity (FEF50)
* Revision of adverse events

4.5 Statistical analysis The study hypothesis will be tested by examining patients´ change from baseline in asthma control (ACT/C-ACT), HR-QoL (PAQLQ/Mini-AQLQ), and in MARS scores between asthma management groups. Results will be summarized between each group as mean scores and analysed by paired t-tests.

4.8 Withdrawal A patient should be withdrawn from the trial if, in the opinion of the investigator, it is medically necessary, or if it is the wish of the patient. In any circumstances the reasons for withdrawal should be documented in the Study termination report. Participants who discontinue from the study for any reason will be replaced.

4.9 Safety

An adverse event (AE) is any untoward medical occurrence in participants using or not using Asthmatuner. AE include the following:

* All suspect adverse reaction
* All reactions from medical overdose, abuse, withdrawal, sensitivity or toxicity
* Apparently unrelated illness, including the worsening of a preexisting illness
* Injury or accident
* Abnormalities in physiological testing or physical examination
* Laboratory abnormalities that require clinical intervention or further investigation unless they are associated with an already reported clinical event.

Preexisting conditions In this trial, a preexisting condition i.e. asthma, should not be reported as an adverse event unless the condition worsens or episodes increases (i.e. exacerbations) in the frequency during the adverse event reporting period.

Procedures Diagnostics and therapeutic non-invasive and invasive procedures, such as surgery, should not be reported as adverse events. However, the medical condition for which the procedure was performed should be reported if it meets the definition of an AE. The AE reporting period begins upon starting the use of Asthmatuner or conventional management (visit 1).

Each participant will be questioned about AE for each visit 2 and 3. All AE that occur in the trial should be reported to investigator and specified in the participants´ medical journal and in a separate AE form with following information:

* Type of AE
* Date and time of AE
* Association with Asthmatuner (No/Yes/Unknown)
* Gravity (Serious or Non-serious)
* Reporting time
* Follow-up (resolved or unresolved)

Gravity

Each AE is to be classified by the investigator as serious or non-serious. This classification of the gravity of the event determines the reporting procedure to be followed. An AE that meets one or more of the following criteria is classified as serious:

* Death
* Life-threatening
* Hospitalization
* Persistent or significant disability/incapacity
* Congenital anomaly/birth defect All serious AE should directly be reported to investigator.

5.0 Ethics The trial will be performed in accordance with the World Medical Assembly Helsinki recommendations guiding physicians in biomedical research involving human subjects [26]. It is the responsibility of the investigators to obtain approval of the trial from regional ethic committee´.

It is the responsibility of the investigators to give each patient prior to inclusion in the trial, full adequate information regarding the trial and the procedures. The patient must be informed about their right to withdraw from the trial at any time. Written patient information must be given to each patient before enrollment. In addition, it is the responsibility of the investigator to obtain signed informed consent from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate is voluntary.
* Age > 6 years
* Diagnosed asthma
* Asthma control score (ACT/C-ACT) less than 20

Exclusion Criteria:

* Ongoing comorbidity affecting the health status of asthma
* Asthma control score (ACT/C-ACT) equal or more than 20
* Participation in other drug trial

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Asthma control | 8 weeks
  Asthma control test
Health-related quality of life | 8 weeks
  Pediatric asthma quality of life questionnaire/Mini-asthma quality of life quest.
Adverse events | 8 weeks
  revision of adverse events

SECONDARY OUTCOMES:
Medical adherence | 8 weeks
  MARS Medicine adherence report scale

CONTACTS AND LOCATIONS:
Locations (1):
- Capio Ringen, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jansson SA, Ronmark E, Forsberg B, Lofgren C, Lindberg A, Lundback B. The economic consequences of asthma among adults in Sweden. Respir Med. 2007 Nov;101(11):2263-70. doi: 10.1016/j.rmed.2007.06.029. Epub 2007 Aug 6. PMID 17689234
- [Background] Brand PL. The clinician's guide on monitoring children with asthma. Paediatr Respir Rev. 2013 Jun;14(2):119-25. doi: 10.1016/j.prrv.2012.07.001. Epub 2012 Aug 24. PMID 23718992
- [Background] Liu WT, Huang CD, Wang CH, Lee KY, Lin SM, Kuo HP. A mobile telephone-based interactive self-care system improves asthma control. Eur Respir J. 2011 Feb;37(2):310-7. doi: 10.1183/09031936.00000810. Epub 2010 Jun 18. PMID 20562122
- [Background] Sadatsafavi M, Rousseau R, Chen W, Zhang W, Lynd L, FitzGerald JM. The preventable burden of productivity loss due to suboptimal asthma control: a population-based study. Chest. 2014 Apr;145(4):787-793. doi: 10.1378/chest.13-1619. PMID 24337140
- [Background] Human D, Crawley F, IJesselmuiden C. Revised declaration of Helsinki. WMA will continue to revise policy as medicine and research changes. BMJ. 2001 Aug 4;323(7307):283-4. No abstract available. PMID 11505938
- [Result] Nordlund B, Konradsen JR, Pedroletti C, Kull I, Hedlin G. The clinical benefit of evaluating health-related quality-of-life in children with problematic severe asthma. Acta Paediatr. 2011 Nov;100(11):1454-60. doi: 10.1111/j.1651-2227.2011.02359.x. Epub 2011 Jun 16. PMID 21595747
- [Result] Fuhrman C, Dubus JC, Marguet C, Delacourt C, Thumerelle C, de Blic J, Delmas MC. Hospitalizations for asthma in children are linked to undertreatment and insufficient asthma education. J Asthma. 2011 Aug;48(6):565-71. doi: 10.3109/02770903.2011.580031. Epub 2011 May 20. PMID 21595608
- [Result] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Result] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Result] Zafari Z, Lynd LD, FitzGerald JM, Sadatsafavi M. Economic and health effect of full adherence to controller therapy in adults with uncontrolled asthma: a simulation study. J Allergy Clin Immunol. 2014 Oct;134(4):908-915.e3. doi: 10.1016/j.jaci.2014.04.009. Epub 2014 May 27. PMID 24875619
- See also: From the Global Strategy for Asthma Management and Prevention, Global Initiative for Asthma (GINA) 2012 — http://www.ginasthma.org/